CLINICAL TRIAL: NCT05623007
Title: Dietary Modulation of Gut Microbiota on Nutritional Status and COVID-19 Infection in Adolescents: Gut-Lung-Axis
Brief Title: Dietary Modulation of Gut Microbiota in Overweight/Obese Adolescents and COVID-19 Infection
Acronym: DIVINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Gadjah Mada University (Other); Universitas Airlangga (Other); University of Melbourne (Other); The Indonesia Endowment Funds for Education, Ministry of Finance Indonesia (Unknown)
Responsible Party: Principal Investigator, Prof Rina Agustina, MD, PhD, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DIVINE
Record Dates: First submitted 2022-10-31; First posted 2022-11-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Health Behavior; Child Development; Adolescent Obesity
Keywords: adolescent; probiotics; COVID-19; overweight; obese
MeSH Terms: conditions — Health Behavior; Pediatric Obesity; COVID-19; Overweight; Obesity | interventions — Probiotics; Exercise

STUDY DESIGN:
Intervention Model Description: The product will be given to 440 overweight/obese adolescents, 220 adolescents as an intervention group, and 220 overweight/obese adolescents as a control group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Enumerator, Investigator, Outcomes Assessor) Participant, enumerator, investigator, and outcomes assessor do not know which one is the intervention product or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 220 overweight/obese adolescents will be given Probiotics and counselling on healthy eating, physical activity, and psychosocial stimulation.
  Interventions: Dietary Supplement: Probiotics; Behavioral: Counselling on healthy eating, physical activity, and psychosocial stimulation
- Control (Placebo Comparator): 220 overweight/obese adolescents will be given placebo probiotics and counselling on healthy eating, physical activity, and psychosocial stimulation.
  Interventions: Behavioral: Counselling on healthy eating, physical activity, and psychosocial stimulation; Dietary Supplement: Placebo probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Combination of 3 probiotic strains: Lactobacillus rhamnosus (LGG), Bifidobacterium animalis subsp. lactis (BB-12), and Lactobacillus acidophilus (LA-5)
  Arms: Intervention
Behavioral: Counselling on healthy eating, physical activity, and psychosocial stimulation — Counselling on healthy eating, physical activity, and psychosocial stimulation.
Dietary Supplement: Placebo probiotics — Maltodextrin
  Arms: Control

SUMMARY:
Probiotic intervention has been currently suggested to provide supportive benefits in promoting health, including alleviating disease symptoms, protecting against diarrhea and respiratory infection, affecting growth and modulating the immune system by improving the beneficial gut microbiota colonization, giving direction on the gut-lung-axis pathway. This indicates that probiotics may become alternative to improve nutrition and reduce the risk of viral infections which may reduce the risk against Severe Acute Respiratory Syndrome Corona Virus-2 (SARS-CoV-2). Introduction to probiotics during adolescence can alleviate inflammation and invert dysbiosis. However, evidence on the effect of probiotic supplementation on enhancing antibody response to SARS COV-2 in adolescents is lacking. Moreover, previous studies showed the potential effect of probiotic supplementation to improve overweight and obesity in adolescents. A bi-directional relationship exists among nutrition, infection, and immunity as changes in one element will affect the others. The main objective of this study is to investigate the effect of dietary modulation of overweight and obese adolescent's gut microbiota through probiotic supplementation combined with healthy eating and physical activity counseling and psychosocial stimulation on nutritional status and antibody response to COVID-19 vaccination. This trial will conduct a 20-week intervention for overweight and obese adolescents.

DETAILED DESCRIPTION:
The adolescence period is the transition from childhood to adulthood. Adolescents are vulnerable to many biomedical exposures, such as a low-quality diet, fewer fruits and vegetable intake, low physical activities, smoking habits, and alcohol consumption; and non-biomedical aspects such as mental depression, parental distress, and household income, which were known to be associated with increased risk of many health outcomes. Obese adolescents are vulnerable to many infections, poor disease outcomes and complications, and lower antibody response to vaccinations. Studies that have investigated Covid-19 incidence in overweight and obese individuals are still scarce. Adolescence is also a sensitive period to microbial change or dysbiosis due to practicing poor diet, low physical activity, inadequate sleep, stress, and substance use (smoking, drugs, and alcohol). Despite the existing prevalence of SARS-COV-2 infections is increasing in adolescents, and the vaccine program is not prioritized in this population, making the prevention strategy for SARS-COV-2 infection may become less effective in this population. Besides, low-quality diet and lifestyle habits and family cluster transmission at home are often not fully addressed in the policy. These factors may be the contributors to the potential highest COVID-19 exposure for children and adolescents. Since exposure among adolescents is linked to serious adverse health effects, effective interventions to improve nutritional outcomes and reduce the risk of COVID-19 infection will provide substantial long-term returns. However, such interventions for adolescents in Indonesia and globally are lacking.

This study is a randomized clinical trial (RCT) and placebo parallel controlled study. The research will be conducted in junior and senior high schools in Jakarta, Surabaya, and Yogyakarta, Indonesia.

In light of COVID-19 outbreak, if face-to-face activities are permitted by (1) national government (Indonesian Ministry of Health), (2) local government (DKI Jakarta), (3) the university, (4) Data Safety Monitoring Board, and (5) by consent of the subject, then the activities need to be strictly adjusted with the COVID-19 prevention measures for both personnel and subjects. All personnel and subjects who will be involved in the activities are required to fill out the COVID-19 symptom screening form prior to the visit and have been vaccinated with a complete dose.

ELIGIBILITY:
Inclusion Criteria:

1. living in Jakarta, Surabaya, and Yogyakarta City for at least 6 months permanently;
2. apparently healthy;
3. male and female, age 12-17 years old;
4. overweight or obese (BMI-for-age z-score >+1SD);
5. have completed at least two dosages of COVID-19 vaccine, the vaccine must be CoronaVac® (Sinovac);
6. minimal 6 months post vaccinated prior to recruitments.
7. parents willing to sign the informed consent and adolescents give informed assent;
8. Must have an active health insurance, for instance BPJS or similar health insurance.

Exclusion Criteria:

1. having a history of COVID-19 infection within the last month confirmed by PCR or antigen from health care facilities or independent laboratory;
2. having a history of chronic and non-communicable diseases, congenital diseases, and disabilities;
3. reported current diagnosed as suspected active Tuberculosis (primary lung TB, miliary TB, bleeding cough bone TB, meningitis TB);
4. having a history of gastrointestinal or malabsorption disorder (such as celiac disease and inflammatory bowel disease) within the last three months or during the study;
5. taking antibiotics during 2 weeks before the start of the study (adolescents will be included after 3 weeks of last antibiotic intake);
6. taking other medications or having diseases that may influence the immune response - i.e. immune deficiencies, immunosuppressants medications, blood transfusion or other blood products;
7. taking insulin and/or anti-dyslipidemia medication;
8. being pregnant and/or breastfeeding.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
BMI-for-age z-scores (BAZ) | 5, 10, 15, and 20 weeks
  Change in BAZ obtain from anthropometric measurements, i.e., weight (kg) and height (m) converted to BMI
Immunoglobulin G (IgG) specific to SARS-COV-2 titer concentrations | 10 and 20 weeks
  Change in IgG specific to SARS-COV-2 titer concentrations assessed by electro chemiluminescence immunoassay (ECLIA)

SECONDARY OUTCOMES:
α-gut microbiota diversity | 20 weeks
  Change in α-diversity measured by 1) Chao1, 2) phylogenetic diversity, and 3) the Shannon index.
β-gut microbiota diversity | 20 weeks
  Change in β -diversity: as the variability in community composition (the identity of taxa observed) among samples
Monoclonal antibody affinity against SARS-COV-2 | 10 and 20 weeks
  Change in equilibrium dissociation constant (KD) of monoclonal antibody against SARS-COV-2 spike protein measured by competitive ELISA
Secretory Immunoglobulin A (sIgA) specific to SARS-COV-2 titer concentrations | 10 and 20 weeks
  Change in sIgA specific to SARS-COV-2 titer concentrations assessed by competitive ELISA
Dietary quality | 5, 10, 15, and 20 weeks
  Change in score of dietary quality assessed by Healthy Eating Index 2015 from 24 hour recalls data

OTHER OUTCOMES:
SARS-COV-2 infection | 20 weeks
  Changes in proportion of symptomatic COVID-19 and positive PCR
Body height | 5, 10, 15, and 20 weeks
  Changes in height-for-age z-score by anthropometric measurement
Abdominal obesity (waist circumference) | 5, 10, 15, and 20 weeks
  Changes in waist circumference by anthropometric measurement
Abdominal obesity (waist-hip ratio) | 5, 10, 15, and 20 weeks
  Changes in waist-hip ratio by anthropometric measurement
Middle upper arm circumference | 5, 10, 15, and 20 weeks
  Changes in middle upper arm circumference by anthropometric measurement
Immunoglobulin M (IgM) against SARS-Cov-2 | 10 and 20 weeks
  Changes in IgM titer concentrations assessed by electro chemiluminescence immunoassay (ECLIA)
Neutralizing antibody against SARS-Cov-2 | 10 and 20 weeks
  Changes in total neutralizing antibody titer assessed by Surrogate Virus Neutralization Test (sVNT)
Gut integrity (zonulin) | 20 weeks
  Changes in the level of serum zonulin assessed by ELISA and Changes in the level of fecal zonulin assessed by ELISA
Gut integrity (occludin) | 20 weeks
  Changes in the level of fecal occludin assessed by ELISA
Gut inflammation | 20 weeks
  Changes in concentration of fecal calprotectin assessed by ELISA
Gut microbiota profiling | 20 weeks
  Changes in composition of gut microbiota assessed by next-generation sequencing (NGS)
Short Chain Fatty Acids (SCFA) | 20 weeks
  Change in concentration of the SCFA by gas chromatograph
Physical activity | 5, 10, 15, and 20 weeks
  Changes in International Physical Activity Questionnaire for Adolescent (IPAQ-A) score, the minimum is 0 metabolic equivalents of task (MET) minutes/week, and the maximum score is 3000 MET minutes/week. Higher score means better outcome.
Body image | 20 weeks
  Changes in Body Shape Questionnaire-34 (BSQ-34) score. The minimum score is 34, and the maximum is 204. Higher score means worse outcome
Depression | 20 weeks
  Changes in Patient Health Questionnaire for Adolescents (PHQ-A) score. The minimum score is 0, and the maximum is 27. Higher scores mean worse outcome.
Self-esteem | 20 weeks
  Changes in Rosenberg Self Esteem Scale. The minimum score is 0, and the maximum score is 37. Higher scores mean better outcome.
Quality of life score | 20 weeks
  Changes in the score of Youth Quality of Life for adolescents-Research version (YQOL-R). The minimum score is 0, and the maximum score is 100. Higher scores mean better outcome.
Morbidity | 5, 10, 15, and 20 weeks
  Type and frequency of illness
Mortality | 5, 10, 15, and 20 weeks
  Type and frequency of illness
Wechsler Intelligence Scale for Children score | 20 weeks
  Changes in Wechsler Intelligence Scale for Children (WISC). The minimum score is 70, and the maximum score is 159. Higher scores mean better outcome.
Brain Derived Neurotropic Factor level | 20 weeks
  Changes in level of Brain Derived Neurotropic Factor (BDNF) assessed by ELISA
Anemia status | 20 weeks
  Changes in hemoglobin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, PhD, Principal Investigator — Dep of Nutrition and Human Nutrition Research Center, IMERI, Fac of Medicine Universitas Indonesia
Locations (1):
- Department of Nutrition (FKUI-RSCM); and Human Nutrition Research Center, Indonesian Medical Education Research Institute (HNRC-IMERI) Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
We will make data from the clinical trials available upon reasonable request subject to approval from the Ministry of Health of the Republic of Indonesia. This will be in accordance with the following regulations: (1) Regulation of the Ministry of Health No. 85 Year 2020 concerning the Transfer and Use of Materials, Information Content, and Data; (2) Law No. 17 Year 2023 on Health; (3) Government Regulation No. 28 Year 2024 on the Implementation Regulation of Law No. 17 of 2023 on Health; (4) Law No. 27 of 2022 on Personal Data Protection. The individual data will be kept anonymous.

REFERENCES:
- [Background] Petta I, Fraussen J, Somers V, Kleinewietfeld M. Interrelation of Diet, Gut Microbiome, and Autoantibody Production. Front Immunol. 2018 Mar 6;9:439. doi: 10.3389/fimmu.2018.00439. eCollection 2018. PMID 29559977
- [Background] Rajput S, Paliwal D, Naithani M, Kothari A, Meena K, Rana S. COVID-19 and Gut Microbiota: A Potential Connection. Indian J Clin Biochem. 2021 Jul;36(3):266-277. doi: 10.1007/s12291-020-00948-9. Epub 2021 Jan 21. PMID 33495676
- [Background] Agustina R, Kok FJ, van de Rest O, Fahmida U, Firmansyah A, Lukito W, Feskens EJ, van den Heuvel EG, Albers R, Bovee-Oudenhoven IM. Randomized trial of probiotics and calcium on diarrhea and respiratory tract infections in Indonesian children. Pediatrics. 2012 May;129(5):e1155-64. doi: 10.1542/peds.2011-1379. Epub 2012 Apr 9. PMID 22492764
- [Background] Abenavoli L, Scarpellini E, Colica C, Boccuto L, Salehi B, Sharifi-Rad J, Aiello V, Romano B, De Lorenzo A, Izzo AA, Capasso R. Gut Microbiota and Obesity: A Role for Probiotics. Nutrients. 2019 Nov 7;11(11):2690. doi: 10.3390/nu11112690. PMID 31703257
- [Derived] Agustina R, Ekawidyani KR, Mutiyani M, Prafiantini E, Nindya TS, Damayanti W, Rejeki PS, Djuari L, Huriyati E, Bines JE, Juffrie M. Study protocol for a randomised controlled trial evaluating the efficacy of dietary modulation of probiotics on nutritional status and antibody response to SARS-CoV-2 in Indonesian adolescents: gut-lung axis (DIVINE). BMJ Open. 2025 Apr 2;15(4):e087934. doi: 10.1136/bmjopen-2024-087934. PMID 40180370